CLINICAL TRIAL: NCT05346666
Title: Possible Immuno-Modulatory Effect of Tocilizumab in Patients With Refractory Status Epilepticus.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other); Principal Investigator Mohanad Omar Ahmed, Msc Pharmacy Practice Department- Horus University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34233/11/20
Record Dates: First submitted 2022-02-24; First posted 2022-04-26 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Phenobarbital; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Group 1 received the conventional treatment for Status Epilepticus including propofol (loading dose is 3 to 5 mg/kg with maintenance of 1 to 15 mg/kg/h), phenobarbital (initial loading dose is 5 to 15 mg/kg over 1 hour. Infusion rates can be maintained at 0.5 to 15 mg/kg/h), and midazolam (a loading dose of 0.2 mg/kg is given with maintenance doses ranging between 0.05 and 2.0 mg/kg/h).
  Interventions: Drug: Tocilizumab Prefilled Syringe [Actemra]. propofole, phenobarbital, midazolam
- Tocilizumab Group (Experimental): Group 2 received the same treatment in group 1 in addition to tocilizumab that was initiated at a dose of 4mg/kg administered twice monthly with 1-week intervals for 3 months. A monthly dose (8mg/kg) of tocilizumab was added if needed.
  Interventions: Drug: Tocilizumab Prefilled Syringe [Actemra]. propofole, phenobarbital, midazolam

INTERVENTIONS:
Drug: Tocilizumab Prefilled Syringe [Actemra]. propofole, phenobarbital, midazolam — Tocilizumab is an immuno-modulatory drug which act as interleukin (IL)-6 receptor inhibitor that blocks IL-6-mediated signal transduction. This drug is known to improve various diseases

SUMMARY:
Recently, the pathogenesis of epilepsy is immuno-modulatory and neuro-inflammatory which is commonly activated in epileptogenic brain regions in humans and is clearly involved in animal models of epilepsy. Inflammatory mediators in the blood and molecular imaging of neuro-inflammation could provide diagnostic, prognostic, and predictive biomarkers for epilepsy, which will be instrumental for patient stratification in future clinical studies. Dysfunction of the blood-brain barrier (BBB) may be responsible for abnormal neuronal firing. Disruption of the BBB causes the leakage of serum protein and leucocyte invasion into the brain. These exogenous inflammatory mediators have the potential to lower seizure thresholds, which could alter channel sensitivity, neurotransmitter uptake or release, and glia-associated regulation of extracellular environments, such as potassium concentration.

ELIGIBILITY:
Inclusion Criteria:

* Age: 15-75 years old.
* Gender: Male and female.
* Newly diagnosed refractory status epilepticus patients who are scheduled to receive anti-epileptic drugs.
* Patients with normal renal and hematological functions.

Exclusion Criteria:

* Old age >75 years old.
* Pregnant or lactating females.
* Severe renal impairment when GFR<30 ml/min.
* Hepatic patients ( not recommended with active hepatic disease or hepatic impairment specially when ALT or AST >3 times ULN).
* Neutropenia when neutrophil count <500 cells/mm3 due to increase the risk of infection.
* Thrombocytopenia when platelet count < 50000 cells/mm3.
* Patients take Immunosuppressant drugs.
* Cancer patient who taking chemotherapy.
* Patients with a known hypersensitivity to any of the used drugs.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
change in the level of inflammatory biomarkers (IL-6, TNF-alpha, IL-1β and NF-κB ) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, Egypt